CLINICAL TRIAL: NCT01677403
Title: A Randomized,Controlled Study to Evaluate the Efficacy,Indications,Adverse Reactions and Resistance of Combined Administration of Nebulized Tobramycin Compared With Systemic Administration Alone in Patients With Bronchiectasis
Brief Title: A Study to Access Safety and Efficacy of Nebulized Tobramycin in Patients With Bronchiectasis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Qi Qian, Principal Investigator, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: qlhqiqian; QL (Registry Identifier: QQian)
Record Dates: First submitted 2012-08-26; First posted 2012-09-03 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Bronchiectasis
Keywords: Bronchiectasis; Tobramycin; nebulised
MeSH Terms: conditions — Bronchiectasis | interventions — Tobramycin; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nebulised Tobramycin (Active Comparator): Nebulised Tobramycin
  Interventions: Drug: Tobramycin
- Nebulised 0.9% Saline (Placebo Comparator): Nebulised 0.9% Saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Tobramycin — Nebulised 80mg twice daily
  Arms: Nebulised Tobramycin
Drug: Saline — Nebulised 5mls 0.9% Saline twice daily
  Arms: Nebulised 0.9% Saline

SUMMARY:
This is a study to evaluate the efficacy,indications,adverse reactions and resistance of combined administration of nebulized tobramycin compared with systemic administration alone in patients with Bronchiectasis in acute exacerbation of Bronchiectasis.

DETAILED DESCRIPTION:
Bronchiectasis is a chronic disorder of the major bronchi and bronchioles characterized by permanent dilation, microbial infection, a persistent inflammatory response with the release of immune mediators and microbial toxins leading to destruction. The origin of bronchiectasis varies, but the presence of microbial infection and a persistent inflammatory response is typical of the disease. The chronic nature of the infection and the associated considerable morbidity provides the rationale for using aerosolized antibiotics for the treatment of bronchiectasis patients.

This is a study of safety and efficacy of combined administration of nebulized tobramycin compared with systemic administration alone in patients with Bronchiectasis in acute exacerbation of Bronchiectasis. Study subjects will be randomized to receive either study drug or placebo by inhalation via a nebulizer. Each subject will complete 14 days of daily dosing.

Clinical laboratory parameters,clinical adverse events and pulmonary function will be evaluated for all study subjects in order to determine the qualitative and quantitative safety and efficacy of nebulized tobramycin.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female study subjects ≥18 years of age and ≤80 years of age
2. Confirmed diagnosis of idiopathic bronchiectasis or postinfectious bronchiectasis
3. Confirmation of infection with P. aeruginosa at screening
4. Are sensitive to Tobramycin
5. Acute exacerbation of bronchiectasis -

Exclusion Criteria:

1. Bronchiectasis due to special causes.
2. Smokers.
3. Are associated with bronchial asthma.
4. Have any serious or active medical or psychiatric illness.
5. Are not tolerant to nebulised tobramycin
6. FEV1.0 reduces ≥ 15% after inhaling tobramycin. -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate change in density of Pseudomonas aeruginosa in sputum | days 1,7,14

SECONDARY OUTCOMES:
To evaluate chang in the amount of sputum | days 1,7,14
To evaluate chang in patients' cough severity | days 1,7,14
To evaluate change in pulmonary function | days 1,7,14

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong University, Jinan, Shandong, China